CLINICAL TRIAL: NCT01944124
Title: A Lifestyle Intervention Supported by Mobile Health Technologies to Improve the Cardiometabolic Risk Profile of Individuals at Risk for Cardiovascular Disease and Type 2 Diabetes.
Brief Title: Exercise and Technology to Reduce Risk in a Rural Population With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); Canadian Diabetes Association (Other)
Responsible Party: Principal Investigator, Rob Petrella, Beryl and Ivey Research Chair, Aging, Rehabilitation and Geriatric Care Research Centre, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 15828
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Metabolic Syndrome X
Keywords: Mobile health; Metabolic syndrome; Exercise prescription; Exercise intervention; Disease prevention; Rural health
MeSH Terms: conditions — Metabolic Syndrome | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Prescription + Mobile Health (Experimental): Received a tailored exercise prescription and mobile health technology kit to track blood pressure, blood glucose, physical activity and body weight.
  Interventions: Behavioral: Mobile Health; Behavioral: Exercise Prescription
- Exercise Prescription (Active Comparator): Received a tailored exercise prescription only.
  Interventions: Behavioral: Exercise Prescription

INTERVENTIONS:
Behavioral: Mobile Health — Participants monitored their blood pressure 3x per week, blood glucose 1x per week, pedometer steps daily and body weight monthly. Measures from devices were transferred or inputted to a smartphone data portal. Planned exercise was logged electronically on the smartphone.
  Arms: Exercise Prescription + Mobile Health
Behavioral: Exercise Prescription — An exercise program was prescribed tailored to participant fitness level (using the Step Test Exercise Prescription (STEP-TM) protocol). Briefly, STEP-TM required participants to step up and down a set of 2 steps 20 times at a comfortable pace. A predictive equation including post-test heart rate, time to complete test, age, body weight and sex was used to calculate fitness. An exercise program was prescribed including aerobic exercise most days of the week for 30-60 minutes in duration at a target heart rate tailored to fitness level. Light resistance training was also prescribed 2-4 times per week.

SUMMARY:
Cardiovascular diseases are the leading cause of death among Canadians. In those with diabetes, cardiovascular complications are responsible for more than 70% of deaths. While there is much interest in identifying and treating risk factors, the exact biological mechanisms, their measurement and optimal ways to prevent and manage them are poorly understood.

Physical activity and regular exercise can prevent diabetes and effectively manage risk factors, but most Canadians do not exercise enough to beneficially manage risk. Tailored exercise prescribed by a family physician has shown promise as a means to increase fitness and reduce risk, but optimal implementation practices remain unknown - especially in rural and remote communities with reduced access to healthcare. Mobile health technologies have proved to be a beneficial tool to achieve blood pressure and blood glucose control in patients with diabetes. These technologies may address the limited access to health interventions in rural and remote regions. However, the potential as a tool to support exercise-based prevention activities unknown.

Therefore, this study was undertaken to investigate the effects of a tailored exercise prescription alone or supported by mobile health technologies to improve cardiovascular risk factors in rural community-dwelling adults at risk for cardiovascular disease and type 2 diabetes.

Adults with cardiovascular risk factors were recruited from rural communities and randomized to either: 1) an intervention group receiving an exercise prescription and devices for monitoring of risk factors with a smartphone data portal equipped with a mobile health application; or 2) an active control group receiving only an exercise prescription.

It was hypothesized that the intervention group would reduce their risk to a greater extent than the active control group following 12 weeks, and that these improvements would be better maintained in the intervention group at 24 and 52 weeks compared to the active control group.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years
* two or more metabolic syndrome risk factors according to National Cholesterol Education Program Adult Treatment Panel III criteria: waist circumference ≥ 88 cm (women) or ≥ 102 cm (men); systolic blood pressure ≥ 135 mmHg and/or diastolic blood pressure ≥ 85 mmHg; fasting plasma glucose ≥ 6.1 mmol/L; triglycerides ≥ 1.7 mmol/L; and high density lipoprotein cholesterol ≤ 1.29 mmol/L (women) or ≤ 1.02 mmol/L (men)

Exclusion Criteria:

* systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110mmHg
* type 1 diabetes
* history of myocardial infarction, angioplasty, coronary artery bypass or cerebrovascular ischemia/stroke
* symptomatic congestive heart failure
* atrial flutter
* unstable angina
* unstable pulmonary disease
* use of medications known to affect heart rate
* second or third degree heart block
* history of alcoholism, drug abuse or other emotional cognitive or psychiatric problems
* pacemaker
* unstable metabolic disease and orthopedic or rheumatologic problems that could impair the ability to exercise

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Petrella, MD, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Gateway Rural Health Research Institute, Seaforth, Ontario, Canada

REFERENCES:
- [Derived] Stuckey MI, Gill DP, Petrella RJ. Does Systolic Blood Pressure Response to Lifestyle Intervention Indicate Metabolic Risk and Health-Related Quality-of-Life Improvement Over 1 Year? J Clin Hypertens (Greenwich). 2015 May;17(5):375-80. doi: 10.1111/jch.12531. Epub 2015 Mar 10. PMID 25757039
- [Derived] Petrella RJ, Stuckey MI, Shapiro S, Gill DP. Mobile health, exercise and metabolic risk: a randomized controlled trial. BMC Public Health. 2014 Oct 18;14:1082. doi: 10.1186/1471-2458-14-1082. PMID 25326074
- [Derived] Stuckey MI, Shapiro S, Gill DP, Petrella RJ. A lifestyle intervention supported by mobile health technologies to improve the cardiometabolic risk profile of individuals at risk for cardiovascular disease and type 2 diabetes: study rationale and protocol. BMC Public Health. 2013 Nov 7;13:1051. doi: 10.1186/1471-2458-13-1051. PMID 24199747